CLINICAL TRIAL: NCT04256317
Title: A Multi-phase, Pharmacokinetics, Safety, and Efficacy Study of ASTX030 (Azacitidine and Cedazuridine) as Monotherapy in Subjects With Myeloid Neoplasm or in Combination With Venetoclax in Subjects With AML (AZTOUND Study)
Brief Title: A Multi-phase Study of ASTX030 (Azacitidine and Cedazuridine) in Myeloid Neoplasm Alone or in Combination With Venetoclax in AML (AZTOUND Study)
Acronym: AZTOUND
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASTX030-01; 2024-515098-93 (Other: EU CT Number)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Myelodysplastic Syndrome/Neoplasm; Chronic Myelomonocytic Leukemia
Keywords: ASTX030; Myeloid Neoplasm; Hematologic Disease; Leukemia; Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); Chronic Myelomonocytic Leukemia (CMML); Vidaza™; Azacitidine; Azacitidine and cedazuridine drug combination; Venetoclax; Venclexta™
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Hematologic Diseases; Leukemia | interventions — Azacitidine; cedazuridine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1 Monotherapy , Stage A (Dose Escalation) (Experimental): In Cycle 1 (28 days per cycle), single dose oral azacitidine will be administered, followed by SC azacitidine, ASTX030 and oral cedazuridine on a specific dosing schedule; in Cycle 2, oral ASTX030 (cedazuridine + azacitidine) will be administered.
  Interventions: Drug: Azacitidine; Drug: ASTX030 (cedazuridine + azacitidine); Drug: Cedazuridine
- Phase 1 Monotherapy, Stage B (Dose Expansion) (Experimental): In Cycle 1 (28 days per cycle), single dose oral azacitidine will be administered, followed by SC azacitidine, ASTX030 and oral cedazuridine on a specific dosing schedule; in Cycle 2, oral ASTX030 (cedazuridine + azacitidine) will be administered. On Day 7 of Cycle 2 drug products will administered in a fed state and all other doses will be administered in fasted state.
  Interventions: Drug: Azacitidine; Drug: ASTX030 (cedazuridine + azacitidine); Drug: Cedazuridine
- Phase 2 Monotherapy, Part B, Sequence A & B (Experimental): In Sequence A: Oral ASTX030 (cedazuridine + azacitidine) will be administered in Cycle 1, followed by SC azacitidine in Cycle 2; all participants will receive ASTX030 in subsequent cycles (Cycles ≥3).
  In Sequence B: SC azacitidine will be administered in Cycle 1, followed by oral cedazuridine + azacitidine tablets/capsules in Cycle 2; all participants will receive ASTX030 in subsequent cycles (Cycles ≥3).
  Interventions: Drug: ASTX030 (cedazuridine + azacitidine); Drug: Azacitidine
- Phase 3 Monotherapy, Sequence A & B (Experimental): In Sequence A: Participants will receive ASTX030 in Cycle 1, followed by SC azacitidine in Cycle 2; all participants will receive ASTX030 in subsequent cycles (Cycles ≥3).
  In Sequence B: Participants will receive SC azacitidine in Cycle 1 followed by ASTX030 in Cycle 2; all participants will receive ASTX030 in subsequent cycles (Cycles ≥3).
  Interventions: Drug: ASTX030 (cedazuridine + azacitidine); Drug: Azacitidine
- Phase 1 Combination Therapy (Experimental): Treatment Arm 1: Participants will receive oral dose of ASTX030 along with ramp-up oral dosing of venetoclax in Cycle 1 (cycle length = 28 days); participants will receive ASTX030 along with venetoclax on a specific dosing schedule in subsequent cycles (Cycles ≥2).
  Treatment Arm 2: Participants will receive SC azacitidine along with ramp-up oral dosing of venetoclax in Cycle 1 (cycle length = 28 days); participants will receive SC azacitidine along with oral dose of venetoclax on a specific dosing schedule in subsequent cycles (Cycles ≥2). At the beginning of Cycle 5, Arm 2 patients may be permitted to cross over to Arm 1.
  Interventions: Drug: ASTX030 (cedazuridine + azacitidine); Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Tablets/Capsules for oral administration and powder for reconstitution to aqueous suspension for SC administration.
  Other Names: Vidaza™ (powder only)
  Arms: Phase 1 Monotherapy , Stage A (Dose Escalation); Phase 1 Monotherapy, Stage B (Dose Expansion)
Drug: ASTX030 (cedazuridine + azacitidine) — FDC Capsules for oral administration.
  Arms: Phase 1 Combination Therapy; Phase 2 Monotherapy, Part B, Sequence A & B; Phase 3 Monotherapy, Sequence A & B
Drug: Azacitidine — Powder for reconstitution to aqueous suspension for SC administration.
  Other Names: Vidaza™ (powder only)
  Arms: Phase 1 Combination Therapy; Phase 2 Monotherapy, Part B, Sequence A & B; Phase 3 Monotherapy, Sequence A & B
Drug: ASTX030 (cedazuridine + azacitidine) — Tablets/Capsules for oral administration.
  Arms: Phase 1 Monotherapy , Stage A (Dose Escalation); Phase 1 Monotherapy, Stage B (Dose Expansion)
Drug: Cedazuridine — Tablets for oral administration.
  Arms: Phase 1 Monotherapy , Stage A (Dose Escalation); Phase 1 Monotherapy, Stage B (Dose Expansion)
Drug: Venetoclax — Oral tablets.
  Other Names: Venclexta™
  Arms: Phase 1 Combination Therapy

SUMMARY:
Study ASTX030-01 is a multi-phase study comprising of Phases 1-3 Monotherapy arms and a Phase 1 Combination Therapy arm Phase 1 Monotherapy consists of an open-label Dose Escalation Stage (Stage A) using multiple cohorts at escalating dose levels of oral cedazuridine and azacitidine (only one study drug will be escalated at a time) followed by a Dose Expansion Stage (Stage B). Phase 2 Monotherapy is a randomized, open-label, crossover study to compare oral ASTX030 to subcutaneous (SC) azacitidine. Phase 3 Monotherapy is a randomized open-label crossover study comparing the final fixed dose of oral ASTX030 to SC azacitidine. Phase 1 Combination Therapy is an open-label, multicenter, randomized, exploratory study comparing ASTX030 and SC azacitidine in combination with venetoclax in participants with AML.

The duration of this multi-phase study is approximately 7 years.

DETAILED DESCRIPTION:
The Phase 1 and Phase 2 Monotherapy arms have completed enrolment. The Phase 3 Monotherapy and Phase 1 Combination Therapy arms are open for enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Phase 2 Monotherapy:

  1. Has Confirmed MDS, CMML, or other MDS/MPN diagnosis who are candidates to receive and benefit from single agent azacitidine and as applicable according to local country approvals and/or local institution standard practice.
* Phase 3 Monotherapy:

  1. Has confirmed MDS or CMML and is a candidate to receive and benefit from single agent azacitidine as applicable according to local country approvals and/or local institution standard practice:

     a) French-American-British myelodysplastic syndrome subtypes: refractory anemia (RA) or refractory anemia with ringed sideroblasts (if accompanied by neutropenia or thrombocytopenia or requiring transfusions), refractory anemia with excess blasts (RAEB), refractory anemia with excess blasts in transformation (RAEB-T), and CMML or MDS with intermediate-2 or high risk MDS according to the International Prognostic Scoring System (IPSS).
  2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
  3. Participants with adequate organ function.
  4. For participants with prior allogeneic stem cell transplant, no evidence of graft-versus-host disease (GVHD).
  5. Participants with no major surgery within 3 weeks before first study treatment.
  6. Participants with no cytotoxic chemotherapy (excluding hydroxyurea) within 4 weeks before first study treatment.
  7. Is able to swallow the number of tablets/capsules required for the treatment assignment within a 10-minute period and tolerate 4 hours of fasting.
  8. Participants with projected life expectancy of at least 12 weeks.
* Phase 1 Combination Therapy:

  1. Has histological confirmation of newly diagnosed AML by World Health Organization (WHO) 2022 criteria.
  2. Participants with projected life expectancy of at least 12 weeks.
  3. Must be considered ineligible for intensive induction chemotherapy defined by the following:

     a. Aged 75 years or older, or b. Aged 18 to 74 years with at least one of the following comorbidities: i. Severe cardiac disorder (e.g., congestive heart failure requiring treatment, ejection fraction ≤50%, or chronic stable angina).

     ii. Severe pulmonary disorder (e.g., diffusing capacity of the lung for carbon monoxide (DLCO) ≤65% or forced expiratory volume in 1 second [FEV1] ≤65%). iii. Creatinine clearance ≥30 mL/min to <45 mL/min. iv. Moderate hepatic impairment with total bilirubin >1.5 to ≤3.0 × upper limit of normal (ULN).

     v. ECOG Performance Status of 2 or 3.
  4. Has an ECOG Performance Status of 0-2 for participants ≥75 years of age or 0-3 for participants 18 to 74 years of age.

Exclusion Criteria:

* All Monotherapy Phases:

  1. Has an active uncontrolled gastric or duodenal ulcer.
  2. Has poor medical risk because of other conditions.
  3. Has known human immunodeficiency virus (HIV) infection.
  4. Is known to be positive for Hepatitis B or C infection.
  5. Has a life-threatening illness.
  6. Has a history of other malignancies prior to study entry, with the exception of adequately treated in situ carcinoma of the breast or cervix uteri; localized basal cell carcinoma or squamous cell carcinoma of the skin; previous malignancy confined and surgically resected or adequately treated and controlled with other modalities; and any early stage malignancy for which no definitive therapy is required.
  7. Participants with MDS/MPN including CMML who have clinical extramedullary disease including clinically palpable hepatomegaly or splenomegaly.
  8. Has previous treatment with more than 1 cycle of decitabine, azacitidine, or guadecitabine (Phases 2 and 3 only).
  9. Has been treated with any investigational drug or therapy within 2 weeks, or 5 half-lives, whichever is longer, before the protocol-defined first dose of study treatment, or ongoing clinically significant adverse events from previous treatment with investigational drug or therapy.
  10. Has a known or suspected hypersensitivity to cedazuridine or azacitidine or any of their excipients.
  11. Cannot discontinue treatment with any drugs that delay gastric emptying such as glucagon-like peptide-1 (GLP-1) and/or gastric inhibitory polypeptide (GIP) agonists in Cycles 1 and 2 of the study.
  12. Has a known or suspected hypersensitivity to cedazuridine or azacitidine or any of their excipients.
* Phase 1 Combination Therapy:

  1. Has a history of MPN including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia with or without BCR-ABL1 translocation, or AML with BCR-ABL1 translocation.
  2. Has the following karyotype abnormalities: t(15;17) or other acute promyelocytic leukemia variants that remain sensitive to all-trans retinoic acid (ATRA) therapy.
  3. Has known active central nervous system involvement from AML.
  4. Has known human immunodeficiency virus (HIV) infection.
  5. Is known to be positive for Hepatitis B or C infection.
  6. Has severe hepatic impairment
  7. Has severe renal impairment
  8. Has a malabsorption syndrome or other condition that precludes enteral route of administration.
  9. Has a cardiovascular disability status of New York Heart Association Class >2.
  10. Has significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular, or pulmonary disease; or any other medical condition that in the opinion of the investigator would adversely affect his/her participation in this study.
  11. Has clinically significant uncontrolled systemic infection requiring therapy (viral, bacterial, or fungal).
  12. Has a history of other malignancies prior to study entry with the exception of adequately treated in situ carcinoma of the breast or cervix uteri; localized basal cell carcinoma or squamous cell carcinoma of the skin; previous malignancy confined and surgically resected (or adequately treated and controlled with other modalities); and any early stage malignancy for which no definitive therapy is required.
  13. Has a WBC count >25,000/ microliters (μL) (hydroxyurea treatment is permitted to meet this criterion).
  14. Has received treatment with any of the following:

      1. A hypomethylating agent (azacitidine or decitabine) or venetoclax, including prior treatment for MDS.
      2. Chimeric Antigen Receptor (CAR)-T cell therapy.
      3. Investigational therapies for MDS or AML.
  15. Cannot discontinue treatment with any of the following:

      1. Prophylactic antifungal therapy with CYP3A inhibitor activity or other concomitant medications with moderate or strong CYP3A inhibitor activity ≥7 days or 5 halflives, whichever is greater, prior to Cycle 1 Day 1 (C1D1).
      2. Drugs that are strong CYP3A or P-gp inhibitors ≥7 days or 5 half-lives, whichever is greater, prior to C1D1.
  16. Cannot avoid concomitant drugs known as moderate or strong CYP3A inducers.
  17. Cannot discontinue treatment with any drugs that delay gastric emptying such as GLP-1 and/or GIP agonists in Cycles 1 and 2 of the study.
  18. Is participating in another research study requiring interventions such as drug therapy or study procedures.
  19. Has a known or suspected hypersensitivity to cedazuridine, azacitidine, venetoclax, or any of their excipients.
  20. Has known significant mental illness or other conditions such as alcohol or other substance abuse or addictions
  21. Consumes grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or starfruit ≤7 days prior to C1D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1, 2 and 3 Monotherapy: Total Cycle Area Under the Curve (AUC) From 0 to 24 Hours (AUC0-24) Exposures | Predose and at multiple timepoints post-dose up to 24 hours
  Ratio of azacitidine total cycle AUC0-24 exposures after oral ASTX030 over SC azacitidine.
Phase 1 Combination Therapy: Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 24 months
Phase 1 Combination Therapy: Complete Response (CR) Rate as Assessed by the Investigator | Up to 24 months
Phase 1 Combination Therapy: AUC0-24 of Venetoclax With ASTX030 | Pre-dose and at multiple timepoints post-dose up to 24 hours on Day 7 (with ASTX030] of Cycle 1
Phase 1 Combination Therapy: AUC0-24 of Venetoclax Without ASTX030 | Pre-dose and at multiple timepoints post-dose up to 24 hours on Day 14 (without ASTX030) of Cycle 1
Phase 1 Combination Therapy: Maximum Plasma Concentration (Cmax) of Venetoclax With ASTX030 | Pre-dose and at multiple timepoints post-dose up to 24 hours on Day 7 (with ASTX030] of Cycle 1
Phase 1 Combination Therapy: Cmax of Venetoclax Without ASTX030 | Pre-dose and at multiple timepoints post-dose up to 24 hours on Day 14 (without ASTX030) of Cycle 1

SECONDARY OUTCOMES:
Phase 1, 2 and 3 Monotherapy: Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 36 months
Phase 1, 2 and 3 Monotherapy: Change in Deoxyribonucleic Acid (DNA) Methylation | Baseline in Phase 1 to the end of Cycle 2 in Phase 3 (28 days per cycle)
  Percent long interspersed nuclear elements 1 (LINE-1) methylation change (demethylation) from baseline in Cycle 1 (Phase 1) and compared between SC azacitidine and ASTX030 in Cycles 1 and 2 (Phase 2 and 3).
Phase 1, 2 and 3 Monotherapy: Best CR Rate in Participants with MDS, CMML, or MDS/Myeloproliferative Neoplasms (MPN) | Up to 36 months
Phase 1, 2 and 3 Monotherapy: AML-free Survival for Participants with MDS, CMML, or MDS/MPN | Up to 36 months
  Number of days from the date of randomization (date of first treatment in Phase 1) to either the date of MDS, CMML, or MDS/MPN progression to AML or the date of death from any cause
Phase 1, 2 and 3 Monotherapy: Duration of Response | Up to 36 months
  Number of days from the date that criteria are met for response until the first date that recurrent or progressive disease is documented by the investigating physician
Phase 1, 2 and 3 Monotherapy: Overall Survival | Up to 36 months
  Number of days from the date the participant was randomized (date of first treatment in Phase 1) to the date of death, regardless of cause
Phase 1, 2 and 3 Monotherapy: Time to Response | Up to 36 months
  Number of days from the start of treatment until the participant's first day of best response
Phase 1, 2 and 3 Monotherapy: Red Blood Cell (RBC) Transfusion Independence (TI) | Up to 36 months
  Number of participants with RBC TI, defined as no RBC transfusion for 56 consecutive days while maintaining hemoglobin ≥8 g/dL
Phase 1, 2 and 3 Monotherapy: Platelet Transfusion Independence (TI) | Up to 36 months
  Number of participants with platelet TI, defined as no platelet transfusion for 56 consecutive days while maintaining platelets ≥20×10^9/L
Phase 1, 2 and 3 Monotherapy: AUC of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose on Days 1, 2 and 7 of Cycle 1 and Cycle 2 (cycle length=28 days)
Phase 1, 2 and 3 Monotherapy: Cmax of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose on Days 1, 2 and 7 of Cycle 1 and Cycle 2 (cycle length=28 days)
Phase 1, 2 and 3 Monotherapy: Time to Reach Cmax (Tmax) of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose on Days 1, 2 and 7 of Cycle 1 and Cycle 2 (cycle length=28 days)
Phase 1B, Food Effect Cohort: AUC of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose on Day 7 of Cycle 2 (cycle length=28 days)
Phase 1B Monotherapy, Food Effect Cohort: Cmax of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose on Day 7 of Cycle 2 (cycle length=28 days)
Phase 1B Monotherapy, Food Effect Cohort: Tmax of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose on Day 7 of Cycle 2 (cycle length=28 days)
Phase 1 Combination Therapy: AUC0-24 of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose up to 24 hours on Day 7 of Cycles 1 and 2 (cycle length = 28 days)
Phase 1 Combination Therapy: Cmax of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose on Day 7 of Cycles 1 and 2 (cycle length = 28 days)
Phase 1 Combination Therapy: Tmax of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose on Day 7 of Cycles 1 and 2 (cycle length = 28 days)
Phase 1 Combination Therapy: AUC0-9 of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose up to 9 hours on Day 7 of Cycles 1 and 2 (cycle length = 28 days)
Phase 1 Combination Therapy: AUC0-inf of Azacitidine, Cedazuridine and Cedazuridine-epimer | Predose and at multiple timepoints post-dose on Day 7 of Cycles 1 and 2 (cycle length = 28 days)
Phase 1 Combination Therapy: AUC of SC Azacitidine and Venetoclax | Predose and at multiple timepoints post-dose on Day 7 of Cycles 1 and 2 (cycle length = 28 days)
Phase 1 Combination Therapy: AUC of Venetoclax, Azacitidine, and Cedazuridine | Predose and at multiple timepoints post-dose on Day 7 of Cycles 1 and 2 (cycle length = 28 days)
Phase 1 Combination Therapy: Cmax of SC Azacitidine and Venetoclax | Predose and at multiple timepoints post-dose on Day 7 of Cycles 1 and 2 (cycle length = 28 days)
Phase 1 Combination Therapy: Cmax of Venetoclax, Azacitidine, and Cedazuridine | Predose and at multiple timepoints post-dose on Day 7 of Cycles 1 and 2 (cycle length = 28 days)
Phase 1 Combination Therapy: Tmax of Venetoclax, Azacitidine, and Cedazuridine | Predose and at multiple timepoints post-dose on Day 7 of Cycles 1 and 2 (cycle length = 28 days)
Phase 1 Combination Therapy: CR and Complete Response with Partial Hematologic Recovery (CRh) Rate | Up to 24 months
Phase 1 Combination Therapy: CR and Complete Response with Incomplete Hematologic Recovery (CRi) Rate | Up to 24 months
Phase 1 Combination Therapy: Time to CR and CRh | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (73):
- United States (25):
  - Keck School of Medicine of USC, Los Angeles, California
  - UC Irvine Health - Chao Family Comprehensive Cancer Center, Orange, California
  - Yale University, New Haven, Connecticut
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Emory - Winship Cancer Institute, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - John Theurer Cancer Center / Hackensack University, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - New York University Langone Hospital - Long Island, Mineola, New York
  - Perlmutter Cancer Center - 34th Street, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Rochester - Wilmot Cancer Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center (OSUCCC) - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Oregon Oncology Specialists, Salem, Oregon
  - Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute dba Baylor Scott & White Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Eastern Health - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Czechia (4):
  - Fakultni Nemocnice Ostrava, Ostrava, Moravian-Silesian
  - Fakultní Nemocnice Královské Vinohrady, Prague, Prague
  - Vseobecna Fakultni Nemocnice v Praze, Prague, Prague
  - Fakultni Nemocnice Brno, Brno, South Moravian
- France (3):
  - Institut Universitaire du Cancer de Toulouse (IUCT) Oncopole, Toulouse, Haute-Garonne
  - Hôpital l'Archet, Nice, Provence-Alpes-Côte d'Azur Region
  - Hôpital Saint-Louis, Paris, Île-de-France Region
- Germany (4):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Städtisches Klinikum Braunschweig, Braunschweig, Lower Saxony
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
- Hungary (4):
  - Szent-Györgyi Albert Klinikai Központ, II. sz. Belgyógyászati Klinika és Kardiológiai Központ, Szeged, Csongrád megye
  - Petz Aladár Győr-Moson-Sopron Vármegyei Egyetemi Oktató Kórház, Győr, Győr-Moson-Sopron
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Semmelweis Egyetem Belgyógyászati és Hematológiai Klinika, Budapest
- Italy (9):
  - Ospedale Santa Maria delle Croci di Ravenna, Ravenna, Emilia-Romagna
  - Azienda Ospedaliero - Universitaria Careggi, Florence, Florence
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino, Turin
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico Sant Orsola-Malpighi, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Fondazione PTV - Policlinico Tor Vergata, Roma
  - Umberto I - Policlinico di Roma, Roma
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino
- Poland (3):
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin, Lublin Voivodeship
  - Wojewódzkie Wielospecjalistyczne Centrum, Lodz, Lódzkie
  - Szpitale Pomorskie Spółka Z Ograniczoną Odpowiedzialnością, Gdynia, Pomeranian Voivodeship
- Spain (16):
  - Institut Català d'Oncologia Badalona, Badalona, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Institut Català d'Oncologia Girona (ICO Girona), Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Clínica Universidad de Navarra - Madrid, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Quirónsalud Málaga, Málaga
  - Complejo Asistencial Universitario de Salamanca - Hospital Clínico, Salamanca
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (3):
  - King's College Hospital NHS Foundation Trust, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - University Hospital Southampton NHS Foundation Trust, Southampton, England

IPD SHARING:
Plan to Share IPD: No